CLINICAL TRIAL: NCT06354907
Title: Improving Mental Health in School-age Children Through the Kids' Empowerment Program (KEP)
Acronym: KEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sandra A Graham-Bermann, Professor of Psychology, College of Literature, Science, and the Arts and Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00150780
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Child Mental Disorder
Keywords: Mental Health; Intervention
MeSH Terms: conditions — Neurodevelopmental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two groups of children and their parent will be compared and evaluated twice (twelve weeks apart). The first group (approximately half of the sample) will participate in the Kids' Empowerment Program in their classroom and their parent will complete assessments online. The second group will complete both assessments and then receive the program in their classroom after the 12 week interval.
Who Masked: Participant
Masking Description: To minimize the possibility of a breach in confidentiality, each child's and parent's information is protected with a code number that will be associated with all of their study materials instead of their name. All identifying information is stored in a separate locked cabinet in the office of Dr. Graham-Bermann. All other study materials (without names) will be kept in a locked cabinet in the research laboratory of Dr. Graham-Bermann to maintain privacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The KEP Group (Experimental): Children in the KEP group will be interviewed before and after participation in the 12 weeks Kids' Empowerment Program in their classroom. Their parent will complete an online assessment via survey software before their child begins the program and again after 12 weeks.
  Interventions: Behavioral: The Kids' Empowerment Program
- The Comparison Group (No Intervention): Children in the comparison group will be interviewed once and again 12 weeks later. Their parent will complete an online assessment once and again 12 weeks later. Children in the Comparison group will then participate in the Kids' Empowerment Program in their classroom.

INTERVENTIONS:
Behavioral: The Kids' Empowerment Program — The 12-session KEP provides support and information while teaching children self-management skills based on techniques derived from a combination of best, evidence-based practices (e.g., using elements of cognitive behavioral therapy, behavioral activation, brief behavioral activation, and interpersonal therapy. Adjustment is enhanced with a comprehensive approach that strengthens cognition (how to think about things), changes behavior (problem solving or planning actions), and focuses on emotions (identifying and expressing feelings), social relationships (peers, parents, siblings), and physical health (de-stressing, exercise). Group leaders follow a training manual with developmentally appropriate scripts, instructions for behavioral applications in (e.g., craft or game activities) and practice plans.
  Arms: The KEP Group

SUMMARY:
Depression and anxiety are major challenges to American children's optimal mental health, with already high rates exacerbated by the Covid-19 pandemic. Yet help is beyond reach for many children who do not have access to care for reasons including a severely depleted cadre of professionally trained service providers, fear of stigma that goes along with a diagnosis, low access to clinics, and lack of insurance. Without help their problems will likely accelerate and become more deleterious to their development as adolescents and young adults. The current study aims to address the lack of care by providing a program in school classrooms that will reduce children's symptoms of depression and anxiety, as well as enhance their emotion regulation and coping skills. The mental health and adjustment of two groups of children are compared and evaluated at twelve week intervals in this clinical trial - those who first participate in the Kids' Empowerment Program (KEP) and a comparison group that participates in the program after the second evaluation. Once proven to be successful, the ultimate goal of the project is to disseminate the program throughout the State of Michigan and beyond, thereby providing children with tools that will empower them to be successful in managing emotional challenges throughout their life.

DETAILED DESCRIPTION:
The aim of this clinical trial is to conduct an evaluation of whether children who participate in the Kids' Empowerment Program (KEP) have fewer symptoms of depression and anxiety after 12 weeks relative to those in the comparison group.

Further, the investigator seeks to identify for whom the program is most helpful and elements of the program that contribute to success. The experimental condition consists of both those who experience the KEP in-person in their classroom (n = 60) and 60 in the comparison condition. Standardized measures assess children's mental health, coping, resilience, and emotion regulation before and after 12 weeks. Those in the comparison group receive the KEP program in their classroom after the second interview. Children are interviewed at school and parents complete an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Child age 6 to 12 years
* Parent consents to participate interviews and the program
* Parent agrees to two assessments

Exclusion Criteria:

* Child age younger than 6 and older than 12
* Child with significant developmental or cognitive delays prohibiting program participation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale | Pre-intervention and 12 weeks later
  Parent reported and child self-rated symptoms of child's anxiety and depression - 25 items, scored 0 to 3, with minimum score of 0 and highest score of 75. Higher scores indicate greater anxiety and depression.
Strengths and Difficulties Questionnaire | Pre-intervention and 12 weeks later
  Parent reported and child self-rated aggression, peer problems, and pro social skills - 15 items (5 items each scale). Scoring ranges from 0 to 2. Minimum score for each scale is 0 and maximum score if 10. Higher scores indicate greater aggression, greater peer problems, and greater prosocial behavior.

SECONDARY OUTCOMES:
Cognitive Emotion Regulation Questionnaire | Pre-intervention and 12 weeks later
  36 items assessing 9 areas of emotion regulation: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination, Positive reappraisal, Putting into perspective, and Catastrophizing. Each subscale consists of 4 items, scored 1 to 4, with a possible range of 4 to 16 for each subscale. Higher scores indicate greater use of that particular emotion regulation strategy.

OTHER OUTCOMES:
EPOCH Questionnaire | Pre-intervention and 12 weeks later
  The 20 item EPOCH is used to measure subjective well-being and includes subscales of Engagement, Perseverance, Optimism, Connectedness, and Happiness. The five subscales consist of 4 items each scored from 1 to 5. The range of scores for each subscale is from 4 to 20. Child self-report and parent report of child. Higher scores indicate greater well-being for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Graham-Bernann, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beck, J. S. (2011), Cognitive behavior therapy: Basics and beyond (2nd ed.), New York, NY: The Guilford Press, pp. 19-20.
- [Result] Cuijpers P, Donker T, Weissman MM, Ravitz P, Cristea IA. Interpersonal Psychotherapy for Mental Health Problems: A Comprehensive Meta-Analysis. Am J Psychiatry. 2016 Jul 1;173(7):680-7. doi: 10.1176/appi.ajp.2015.15091141. Epub 2016 Apr 1. PMID 27032627
- [Result] Funderburk JS, Pigeon WR, Shepardson RL, Maisto SA. Brief behavioral activation intervention for depressive symptoms: Patient satisfaction, acceptability, engagement, and treatment response. Psychol Serv. 2020 Nov;17(4):443-451. doi: 10.1037/ser0000328. Epub 2019 Feb 4. PMID 30714752
- [Result] Mazzucchelli, T. G. (2016). Behavioural activation: Current practice, new applications, and future directions. Clinical Psychologist, 20(1), 3-4. https://doi.org/10.1111/cp.12089
- [Result] Garnefski, Nadia, & Kraaij, V. (2007). The Cognitive Emotion Regulation Questionnaire. European Journal of Psychological Assessment, 23(3), 141-149. doi:10.1027/1015-5759.23.3.141
- [Result] Kern ML, Benson L, Steinberg EA, Steinberg L. The EPOCH Measure of Adolescent Well-Being. Psychol Assess. 2016 May;28(5):586-97. doi: 10.1037/pas0000201. Epub 2015 Aug 24. PMID 26302102
- [Result] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702